CLINICAL TRIAL: NCT06667466
Title: Prospective, Multicenter, Randomized Controlled Trial of Super Pulse Thulium Fiber Laser Combined With Flexible Negative Pressure Suction Sheath Versus Conventional Sheath for the Treatment of Kidney Stones
Brief Title: New Laser and Suction Sheath for Kidney Stone Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yi Shao, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: IIT2024-148
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Kidney Calculi; Ureteral Calculi
MeSH Terms: conditions — Kidney Calculi; Ureteral Calculi | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sTFL + Flexible Negative-Pressure UAS: Under general anesthesia, a guidewire is first inserted. Then, the Flexible Negative Pressure UAS is inserted along the guidewire to the stone site. A ureteroscope is inserted through the sheath to the stone site. The sTFL is used to fragment the stone with a power setting of 0.8J and a frequency of 12 - 20Hz. Simultaneously, the fragmented stones are removed by negative pressure suction.
  Interventions: Device: Super Pulsed Thulium Fiber Laser (sTFL) + Flexible Negative Pressure Ureteral Access Sheath (UAS) Intervention
- sTFL + Conventional UAS: Under general anesthesia, the Conventional UAS is inserted to the upper ureter or the ureteropelvic junction. A ureteroscope is inserted through the sheath to the stone site. The sTFT is used to fragment the stone with a power setting of 0.8J and a frequency of 12 - 20Hz. After fragmentation, the stones are removed by a stone basket.
  Interventions: Device: Super Pulsed Thulium Fiber Laser (sTFL) + Conventional Ureteral Access Sheath (UAS) Intervention

INTERVENTIONS:
Device: Super Pulsed Thulium Fiber Laser (sTFL) + Flexible Negative Pressure Ureteral Access Sheath (UAS) Intervention — The intervention combines a Super Pulsed Thulium Fiber Laser (sTFL) with a power setting of 0.8J and a frequency of 12 - 20Hz for stone fragmentation and a Flexible Negative Pressure Ureteral Access Sheath (UAS) that allows access to the stone site and enables negative pressure suction for stone removal.
  Groups: sTFL + Flexible Negative-Pressure UAS
Device: Super Pulsed Thulium Fiber Laser (sTFL) + Conventional Ureteral Access Sheath (UAS) Intervention — The intervention combines a Super Pulsed Thulium Fiber Laser (sTFL) with a power setting of 0.8J and a frequency of 12 - 20Hz for stone fragmentation and a Conventional Ureteral Access Sheath (UAS) used for access to the upper ureter or ureteropelvic junction for stone treatment.
  Groups: sTFL + Conventional UAS

SUMMARY:
The goal of this clinical trial is to learn if the combination of super pulsed thulium fiber laser (sTFL) with a flexible negative pressure suction sheath is more effective and safer than sTFL with a conventional sheath in treating kidney stones and/or ureteral stones. The main questions it aims to answer are:

Does the sTFL with a flexible negative pressure suction sheath have a higher stone - free rate than the sTFL with a conventional sheath? Does the sTFL with a flexible negative pressure suction sheath have fewer complications than the sTFL with a conventional sheath?

Researchers will compare the two treatment groups to see if there are differences in stone - free rate and complication rates.

Participants will:

Undergo ureteroscopic lithotripsy surgery. In the experimental group, have a flexible negative pressure suction sheath inserted along a guidewire to the stone site under general anesthesia, then have a ureteroscope inserted through the sheath to the stone site, and have the stone fragmented by sTFL with a power setting of 0.8J and a frequency of 12 - 20Hz while the fragments are removed by negative pressure suction.

In the control group, have a conventional sheath inserted to the upper ureter or the ureteropelvic junction under general anesthesia, then have a ureteroscope inserted through the sheath to the stone site, and have the stone fragmented by sTFL with a power setting of 0.8J and a frequency of 12 - 20Hz and the fragments removed by a stone basket.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, controlled clinical trial aimed at comparing the efficacy and safety of super pulsed thulium fiber laser (sTFL) combined with a flexible negative pressure suction sheath versus sTFL combined with a conventional sheath in the treatment of kidney stones and/or ureteral stones.

1. Background and Rationale Urinary calculi are common, with a significant recurrence rate. Incomplete stone removal during treatment is a contributing factor to recurrence. The flexible negative pressure suction sheath offers potential advantages over the conventional sheath, and when combined with the high-performance sTFL, may provide better treatment outcomes. However, a clinical comparison of these combinations has been lacking.
2. Study Design

   Multicenter: Involving hospitals such as Shanghai Jiao Tong University School of Medicine Affiliated First People's Hospital, Shanghai Jiao Tong University School of Medicine Affiliated Sixth People's Hospital, Shanghai Jiao Tong University School of Medicine Affiliated Ninth People's Hospital, and Weifang Hospital of Traditional Chinese Medicine.

   Randomization: Simple randomization is used, with a 1:1 ratio of participants assigned to the experimental group (sTFL + flexible negative pressure suction sheath) and the control group (sTFL + conventional sheath) via a central randomization system.

   Blinding: A third-party independent assessment method is employed. Two radiologists blinded to the patient's group and clinical information will evaluate the CT scans at 3 months postoperatively to determine the stone - free rate.
3. Participants

   Inclusion Criteria: Adults aged 18 years or older, diagnosed with kidney stones and/or ureteral stones with a diameter between 6mm and 20mm, scheduled for ureteroscopic lithotripsy (fURS) under general anesthesia, with a negative preoperative urine culture, and having provided informed consent.

   Exclusion Criteria: Isolated kidney, history of kidney transplant or urinary diversion surgery, congenital urinary tract anomalies, coagulation disorders, severe cardiac or pulmonary diseases, malignant tumors, immunodeficiency, neurogenic bladder, inability to provide informed consent, untreated urinary tract infection, known anatomical abnormalities preventing sheath access to the stone or relevant sites, pregnancy, and those who cannot be treated under the specified anesthesia methods.
4. Interventions

   Experimental Group: Under general anesthesia, a flexible negative pressure suction sheath is inserted along a guidewire to the stone site, followed by insertion of a ureteroscope through the sheath to the stone site. The sTFL is used to fragment the stone with a power setting of 0.8J and a frequency of 12 - 20Hz, while the fragments are removed by negative pressure suction.

   Control Group: Under general anesthesia, a conventional sheath is inserted to the upper ureter or the ureteropelvic junction, followed by insertion of a ureteroscope through the sheath to the stone site. The sTFL is used to fragment the stone with a power setting of 0.8J and a frequency of 12 - 20Hz, and the fragments are removed by a stone basket.
5. Outcome Measures

   Primary Outcome Measure: Stone - free rate (SFR), evaluated by non - contrast CT scan at 3 months postoperatively, defined as residual stone diameter < 2mm.

   Secondary Outcome Measures: Surgery time, complication rates (including intraoperative and postoperative complications such as infection, bleeding, and instrument - related injuries), and changes in vital signs (temperature, pulse, respiration, blood pressure).
6. Safety Assessment

   Adverse Events (AE) and Serious Adverse Events (SAE): All AEs and SAEs are monitored, recorded, and reported. AE details include name, occurrence and resolution dates, severity, impact on the study, relationship to the study, measures taken, and outcome. SAEs must be reported to the ethics committee within 24 hours.

   Vital Signs Monitoring: Vital signs are monitored before, during, and within 24 hours after surgery.

   Complication Assessment: Postoperative complications are assessed using the Clavien - Dindo grading system.
7. Sample Size Calculation Based on an assumed superiority of the experimental treatment, with a clinically significant difference in SFR of 5% between the two groups, a sample size of 67 participants per group (considering a 20% dropout rate) was calculated, totaling 134 participants, and the study aims to recruit 140 participants.
8. Data Analysis Descriptive statistics (means and standard deviations for continuous variables, frequencies and percentages for categorical variables) and comparison tests (t - test for continuous variables, Fisher's exact test for categorical variables) will be used. All analyses will be performed using R software version 4.3, with a significance level of P < 0.05.
9. Follow - up Plan

Baseline Visit (Screening Period): Assess potential participants for eligibility, including collecting demographic data, medical history, measuring vital signs, and performing a CT scan.

Intraoperative Visit (Treatment Period): Record surgery time, instrument usage, and monitor vital signs and complications.

Postoperative 24 - hour Visit (Treatment Period): Monitor vital signs, ask about symptoms, and check for complications.

Postoperative 90 - day Visit (Follow - up Period): Evaluate stone clearance by CT scan and assess symptom recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Diagnosed with kidney stones and/or ureteral stones, and stone diameter is ≥6mm and ≤20mm
* Plan to undergo fURS lithotripsy
* General anesthesia to complete the operation
* The latest urine culture before surgery is negative
* Signed and dated informed consent

Exclusion Criteria:

* Isolated kidney
* Previous history of kidney transplantation or urinary diversion surgery
* Congenital malformations of urinary system
* Abnormal coagulation mechanism due to blood system diseases, liver diseases, etc
* Severe heart or lung disease, malignancy and immune deficiency status
* Neurogenic bladder
* Failure to provide informed consent
* Have an untreated urinary tract infection
* The presence of known anatomic abnormalities (such as ureteral stenosis), urothelial tumors, or stones that can be removed directly without the use of laser lithotripsy
* Pregnant women
* In cases where the stone cannot be reached with a bendable negative pressure suction sheath, or in cases where the stone cannot be reached with a conventional sheath or the pyeloureteral junction
* Epidural anesthesia or lumbar anesthesia to complete the operation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-70 years who plan to undergo ureteral soft endoscopic (fURS) lithotripsy for kidney stones and/or ureteral stones (6-20mm)
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2026-11-20 (Estimated); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | 3 months postoperatively
  The proportion of patients with no residual stone or with residual stone diameter less than 2mm, as determined by non - contrast CT scan. This measure is used to evaluate the effectiveness of the two treatment methods in completely removing the stones.

SECONDARY OUTCOMES:
time of operation | During the surgical procedure
  The incidence of intraoperative and postoperative complications including infection, bleeding, and instrument - related injuries. This helps to evaluate the safety of the two treatment methods
Complication | During the surgical procedure and within 24 hours after the surgical procedure
  The incidence of intraoperative and postoperative complications including infection, bleeding, and instrument - related injuries. This helps to evaluate the safety of the two treatment methods.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Shao, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine